CLINICAL TRIAL: NCT02867020
Title: Phase II Randomized Study of Abiraterone Acetate Plus ADT Versus APALUTAMIDE Versus Abiraterone and APALUTAMIDE in Patients With Advanced Prostate Cancer With Non-castrate Testosterone Levels
Brief Title: Study of Abiraterone Acetate Plus ADT Versus APALUTAMIDE Versus Abiraterone and APALUTAMIDE in Patients With Advanced Prostate Cancer With Non-castrate Testosterone Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Latin American Cooperative Oncology Group (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LACOG 0415
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
Keywords: apalutamide; abiraterone; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; abiraterone; Goserelin; Prednisone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Abiraterone acetate + Prednisone + ADT (Goserelin) (Active Comparator): * Abiraterone administered at a single 1000 mg daily oral dose (4 x 250-mg tablets)
  * Prednisone administered at a 5 mg twice daily oral dose
  * Goserelin administered as subcutaneous injections of 10.8mg every 3 months
  Interventions: Drug: Apalutamide; Drug: Abiraterone; Drug: ADT
- APALUTAMIDE monotherapy (Experimental): o APALUTAMIDE administered at a single 240 mg daily oral dose (4 x 60 mg tablets)
  Interventions: Drug: Apalutamide
- Abiraterone acetate + Prednisone + APALUTAMIDE (Experimental): * Abiraterone administered at a single 1000 mg daily oral dose (4 x 250 mg tablets)
  * Prednisone administered at a 5 mg twice daily oral dose
  * APALUTAMIDE administered at a single 240 mg daily oral dose (4 x 60 mg tablets)
  Interventions: Drug: Apalutamide; Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: Apalutamide — APALUTAMIDE 240-mg orally once daily (4 x 60-mg tablets) will be administered on a continual basis. For the purpose of scheduling the study assessments and treatment compliance a treatment cycle is defined as 28 days.
Drug: Abiraterone — Abiraterone acetate 1,000 mg (four 250 mg tablets) should be taken orally once daily, in combination with oral dose prednisone 5mg twice daily continuously. For the purpose of scheduling the study assessments and treatment compliance a treatment cycle is defined as 28 days
  Arms: Abiraterone acetate + Prednisone + ADT (Goserelin); Abiraterone acetate + Prednisone + APALUTAMIDE
Drug: ADT — Dosing of goserelin (dose and frequency of administration) will be consistent with the prescribing information and should only be adjusted if clinically indicated to achieve and maintain subcastrate concentrations of testosterone (50 ng/dL or 1.7 nM).
  Other Names: Goserelin
  Arms: Abiraterone acetate + Prednisone + ADT (Goserelin)
Drug: Prednisone — Subjects will receive prednisone 10mg/day.
  Arms: Abiraterone acetate + Prednisone + APALUTAMIDE

SUMMARY:
Evaluation of the activity, safety and patients reported outcome of ADT plus abiraterone, abiraterone plus APALUTAMIDE (a second-generation antiandrogen) or APALUTAMIDE alone in hormone naïve locally advanced or metastatic prostate cancer which ADT was indicated.

DETAILED DESCRIPTION:
Based on the current guidelines, ADT alone or combined with is antiandrogens are considered the appropriate active therapy for the patient population planned for this study. Recent data showed that chemotherapy also benefit patients in this setting. Even though, there is a clear unmet medical need for alternative treatment option in metastatic hormone sensitive prostate cancer (mHSPC). Treatments that can delay disease progression, and are associated with less comorbidities would be of significant clinical benefit in this patient population. The study is designed to assess the efficacy and safety of abiraterone plus APALUTAMIDE (a second-generation antiandrogen) or APALUTAMIDE alone without castration side effects and the other arm a combination of ADT and abiraterone; this last arm is to reflect an Abiraterone ongoing pivotal trial (LATITUDE), that assess the efficacy of adding abiraterone to castration in this setting of patients. Abiraterone had already showed clinical benefit in CRPC patients without prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate adenocarcinoma;
2. Hormone naïve patients with indication to ADT in the following settings:

   * Advanced loco-regional disease not amenable to curative local therapy (surgery or radiotherapy): T category T3/4 or node positive
   * Biochemical relapse after primary treatment (surgery or radiotherapy): patients in whom primary therapy is not appropriate or feasible with Previously treated with radical surgery and/or radiotherapy, now relapsing with at least one of the criteria: PSA >= 4 ng/ml and rising with doubling time less than 10 months. or PSA >= 20 ng/ml or N+ or M+
   * Newly diagnosed metastatic disease: Tany Nany M+
3. Patient is asymptomatic or moderately symptomatic regarding bone symptoms, i.e., no need for palliative radiation or radionuclide therapy;
4. Non-castration level of testosterone > 230ng/dL (> 8 nmol/L);
5. Baseline level of prostatespecific antigen (PSA) > 2ng/dL;
6. ECOG performance status of 0 to 2;
7. Adequate hematologic, hepatic and renal function:

   1. hemoglobin > 10 g/dL, neutrophils > 1.5×109 / L, platelets> 100×109 / L;
   2. total bilirubin < 1.5x upper limit of normal (ULN); alanine (ALT) and aspartate (AST) aminotransferase < 2.5 x ULN;
   3. serum creatinine < 1.5x ULN; potassium > 3.5 mM;
8. No previous cancer (except treated basal-cell skin cancer);
9. Written informed consent obtained prior to any study procedure;
10. Men age 18 years and older;
11. Agrees to use a condom and another effective method of birth control if he is having sex with a woman of childbearing potential or agrees to use a condom if he is having sex with a woman who is pregnant.

Exclusion Criteria:

1. Prostate adenocarcinoma with neuroendocrine differentiation or small cell histology;
2. Biochemical recurrence without evidence of clinical or radiological disease;
3. Use of hormonal therapy or chemotherapy prior to randomization. Exception is courses of hormone therapy for localised disease must have been completed at least 12 months previously. It can have been given as adjuvant or neoadjuvant therapy.
4. Prior radiation therapy for a primary tumour within the 3 months before enrollment or for the treatment of metastases;
5. Known or suspected brain or skull metastases or leptomeningeal metastatic disease;
6. Any concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study;
7. Administration of an investigational therapeutic or invasive surgical procedure (not including surgical castration) within 28 days of Cycle 1 Day 1 or currently enrolled in an investigational study;
8. Active or symptomatic viral hepatitis or chronic liver disease; ascites or bleeding disorders secondary to hepatic dysfunction;
9. Current or prior treatment with anti-epileptic medications for the treatment of seizures;
10. Impaired cardiac function, including any of the following:

    1. Uncontrolled hypertension (systolic blood pressure ≥160 mmHg or diastolic BP ≥95 mmHg);
    2. Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events or history of cardiac failure in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class II-IV heart disease;
    3. Existing atrial fibrillation with or without pharmacotherapy. Other cardiac arrhythmia requiring pharmacotherapy;
    4. History of seizure or condition that may predispose to seizure (including, but not limited to prior stroke, transient ischemic attack or loss of consciousness ≤1 year prior to randomization; brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect);
11. Specific underlying conditions for oral agents. For example: impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of abiraterone or APALUTAMIDE (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
12. General excluded medications (e.g., relevant to cytochrome P450 interactions)

    1. Use of prescription drugs within 14 days prior to dosing or over-the-counter (OTC) medication within 7 days prior to dosing;
    2. Consumption of grapefruit product or St John's wort within 7 days prior to dosing;
    3. G-CSF, GM-CSF, erythropoietin, etc;
    4. Coumadin;
    5. Drugs which may cause QT prolongation;
    6. Known sensitivity to drugs or metabolites from similar classes;
    7. Known or suspected contraindications or hypersensitivity to APALUTAMIDE, bicalutamide or GnRH agonists or any of the components of the formulations;
13. Any condition or situation which, in the opinion of the investigator, would put the subject at risk, may confound study results, or interfere with the subject's participation in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients that achieves an undetectable PSA level, defined as ≤ 0.2 ng/mL | Week 25

SECONDARY OUTCOMES:
PSA progression rate | Week 25
  Determination of PSA progression rate among the three experimental arms
Comparison of PSA progression rate | Week 25
  Comparison of PSA progression rate among the three experimental arms
PSA response of 50 and 80% | Week 25
  Determination of PSA response of 50 and 80% among the three experimental arms
Comparison of PSA response of 50 and 80% | Week 25
  Comparison of PSA response of 50 and 80% among the three experimental arms
Maximum PSA declines | Baseline up to week 25 to 52
  Determination of maximum PSA declines among the three experimental arms
Overall PSA change | Baseline up to week 25 to 52
  Determination of overall PSA change among the three experimental arms
Hormonal levels during treatment | Baseline up to week 25
Comparison of hormonal levels during treatment | Baseline up to week 25
  Comparison of hormonal levels during treatment among the three experimental arms
Evaluation of bone mineral density according to RECIST 1.1 | Week 25
Comparison of bone mineral density according to RECIST 1.1 between three experimental groups | Week 25
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Baseline to 2 years of follow-up
Number of participants with pain progression assessed by BPI-SF of three experimental arms | Baseline up to week 25
Number of participants in opioid use during treatment among three experimental arms | Baseline up to week 25
Comparison of pain progression assessed by opioid use | Baseline up to week 25
  Comparison of pain progression assessed by opioid use between the experimental arms
Comparison of pain progression assessed by BPI-SF questionnaire | Baseline up to week 25
  Comparison of pain progression assessed by BPI-SF between the experimental arms
Quality of life assessed by FACT-P questionnaire | Baseline up to week 25
  Quality of life assessed by FACT-P questionnaire of the experimental arms
Comparison of quality of life assessed by FACT-P questionnaire | Baseline up to week 25
  Comparison of quality of life assessed by FACT-P questionnaire between the experimental arms
Radiographic progression-free survival (rPFS) | Week 25
  Radiographic progression-free survival (rPFS) among the experimental arms

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Maluf, MD, Principal Investigator — Beneficiência Portuguesa de São Paulo; Gustavo Werutsky, MD, Study Director — Latin American Cooperative Oncology Group
Locations (14):
- Brazil (14):
  - CRIO, Fortaleza, Ceará
  - Clínica AMO, Salvador, Estado de Bahia
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Oncologia Rede D'Or S.A., Rio de Janeiro, Rio de Janeiro
  - Liga Norte Riograndense de Oncologia, Natal, Rio Grande do Norte
  - Hospital de Caridade de Ijuí, Ijuí, Rio Grande do Sul
  - CPO - Pucrs, Porto Alegre, Rio Grande do Sul
  - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Centro de Pesquisa Clínica em Hematologia e Oncologia - CEPHO, Santo André, São Paulo
  - Grupo COI, Rio de Janeiro
  - Beneficiencia Portuguesa de São Paulo/Hospital São José, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - IBCC, São Paulo
  - ICESP, São Paulo

REFERENCES:
- [Background] Hershman DL, Unger JM, Wright JD, Ramsey S, Till C, Tangen CM, Barlow WE, Blanke C, Thompson IM, Hussain M. Adverse Health Events Following Intermittent and Continuous Androgen Deprivation in Patients With Metastatic Prostate Cancer. JAMA Oncol. 2016 Apr;2(4):453-61. doi: 10.1001/jamaoncol.2015.4655. PMID 26720308
- [Background] Rozet F, Roumeguere T, Spahn M, Beyersdorff D, Hammerer P. Non-metastatic castrate-resistant prostate cancer: a call for improved guidance on clinical management. World J Urol. 2016 Nov;34(11):1505-1513. doi: 10.1007/s00345-016-1803-9. Epub 2016 Mar 17. PMID 26988552
- [Background] Crawford ED, Higano CS, Shore ND, Hussain M, Petrylak DP. Treating Patients with Metastatic Castration Resistant Prostate Cancer: A Comprehensive Review of Available Therapies. J Urol. 2015 Dec;194(6):1537-47. doi: 10.1016/j.juro.2015.06.106. Epub 2015 Jul 18. PMID 26196735
- [Background] Gartrell BA, Coleman R, Efstathiou E, Fizazi K, Logothetis CJ, Smith MR, Sonpavde G, Sartor O, Saad F. Metastatic Prostate Cancer and the Bone: Significance and Therapeutic Options. Eur Urol. 2015 Nov;68(5):850-8. doi: 10.1016/j.eururo.2015.06.039. Epub 2015 Jul 4. PMID 26153564
- [Background] Barrie SE, Potter GA, Goddard PM, Haynes BP, Dowsett M, Jarman M. Pharmacology of novel steroidal inhibitors of cytochrome P450(17) alpha (17 alpha-hydroxylase/C17-20 lyase). J Steroid Biochem Mol Biol. 1994 Sep;50(5-6):267-73. doi: 10.1016/0960-0760(94)90131-7. PMID 7918112
- [Background] Attard G, Reid AH, A'Hern R, Parker C, Oommen NB, Folkerd E, Messiou C, Molife LR, Maier G, Thompson E, Olmos D, Sinha R, Lee G, Dowsett M, Kaye SB, Dearnaley D, Kheoh T, Molina A, de Bono JS. Selective inhibition of CYP17 with abiraterone acetate is highly active in the treatment of castration-resistant prostate cancer. J Clin Oncol. 2009 Aug 10;27(23):3742-8. doi: 10.1200/JCO.2008.20.0642. Epub 2009 May 26. PMID 19470933
- [Background] Attard G, Reid AH, Yap TA, Raynaud F, Dowsett M, Settatree S, Barrett M, Parker C, Martins V, Folkerd E, Clark J, Cooper CS, Kaye SB, Dearnaley D, Lee G, de Bono JS. Phase I clinical trial of a selective inhibitor of CYP17, abiraterone acetate, confirms that castration-resistant prostate cancer commonly remains hormone driven. J Clin Oncol. 2008 Oct 1;26(28):4563-71. doi: 10.1200/JCO.2007.15.9749. Epub 2008 Jul 21. PMID 18645193
- [Background] Danila DC, Morris MJ, de Bono JS, Ryan CJ, Denmeade SR, Smith MR, Taplin ME, Bubley GJ, Kheoh T, Haqq C, Molina A, Anand A, Koscuiszka M, Larson SM, Schwartz LH, Fleisher M, Scher HI. Phase II multicenter study of abiraterone acetate plus prednisone therapy in patients with docetaxel-treated castration-resistant prostate cancer. J Clin Oncol. 2010 Mar 20;28(9):1496-501. doi: 10.1200/JCO.2009.25.9259. Epub 2010 Feb 16. PMID 20159814
- [Background] O'Donnell A, Judson I, Dowsett M, Raynaud F, Dearnaley D, Mason M, Harland S, Robbins A, Halbert G, Nutley B, Jarman M. Hormonal impact of the 17alpha-hydroxylase/C(17,20)-lyase inhibitor abiraterone acetate (CB7630) in patients with prostate cancer. Br J Cancer. 2004 Jun 14;90(12):2317-25. doi: 10.1038/sj.bjc.6601879. PMID 15150570
- [Background] Reid AH, Attard G, Danila DC, Oommen NB, Olmos D, Fong PC, Molife LR, Hunt J, Messiou C, Parker C, Dearnaley D, Swennenhuis JF, Terstappen LW, Lee G, Kheoh T, Molina A, Ryan CJ, Small E, Scher HI, de Bono JS. Significant and sustained antitumor activity in post-docetaxel, castration-resistant prostate cancer with the CYP17 inhibitor abiraterone acetate. J Clin Oncol. 2010 Mar 20;28(9):1489-95. doi: 10.1200/JCO.2009.24.6819. Epub 2010 Feb 16. PMID 20159823
- [Background] Ryan CJ, Shah S, Efstathiou E, Smith MR, Taplin ME, Bubley GJ, Logothetis CJ, Kheoh T, Kilian C, Haqq CM, Molina A, Small EJ. Phase II study of abiraterone acetate in chemotherapy-naive metastatic castration-resistant prostate cancer displaying bone flare discordant with serologic response. Clin Cancer Res. 2011 Jul 15;17(14):4854-61. doi: 10.1158/1078-0432.CCR-11-0815. Epub 2011 Jun 1. PMID 21632851
- [Background] Ryan CJ, Smith MR, Fong L, Rosenberg JE, Kantoff P, Raynaud F, Martins V, Lee G, Kheoh T, Kim J, Molina A, Small EJ. Phase I clinical trial of the CYP17 inhibitor abiraterone acetate demonstrating clinical activity in patients with castration-resistant prostate cancer who received prior ketoconazole therapy. J Clin Oncol. 2010 Mar 20;28(9):1481-8. doi: 10.1200/JCO.2009.24.1281. Epub 2010 Feb 16. PMID 20159824
- [Background] de Bono JS, Logothetis CJ, Molina A, Fizazi K, North S, Chu L, Chi KN, Jones RJ, Goodman OB Jr, Saad F, Staffurth JN, Mainwaring P, Harland S, Flaig TW, Hutson TE, Cheng T, Patterson H, Hainsworth JD, Ryan CJ, Sternberg CN, Ellard SL, Flechon A, Saleh M, Scholz M, Efstathiou E, Zivi A, Bianchini D, Loriot Y, Chieffo N, Kheoh T, Haqq CM, Scher HI; COU-AA-301 Investigators. Abiraterone and increased survival in metastatic prostate cancer. N Engl J Med. 2011 May 26;364(21):1995-2005. doi: 10.1056/NEJMoa1014618. PMID 21612468
- [Background] Fizazi K, Scher HI, Molina A, Logothetis CJ, Chi KN, Jones RJ, Staffurth JN, North S, Vogelzang NJ, Saad F, Mainwaring P, Harland S, Goodman OB Jr, Sternberg CN, Li JH, Kheoh T, Haqq CM, de Bono JS; COU-AA-301 Investigators. Abiraterone acetate for treatment of metastatic castration-resistant prostate cancer: final overall survival analysis of the COU-AA-301 randomised, double-blind, placebo-controlled phase 3 study. Lancet Oncol. 2012 Oct;13(10):983-92. doi: 10.1016/S1470-2045(12)70379-0. Epub 2012 Sep 18. PMID 22995653
- [Background] Ryan CJ, Smith MR, de Bono JS, Molina A, Logothetis CJ, de Souza P, Fizazi K, Mainwaring P, Piulats JM, Ng S, Carles J, Mulders PF, Basch E, Small EJ, Saad F, Schrijvers D, Van Poppel H, Mukherjee SD, Suttmann H, Gerritsen WR, Flaig TW, George DJ, Yu EY, Efstathiou E, Pantuck A, Winquist E, Higano CS, Taplin ME, Park Y, Kheoh T, Griffin T, Scher HI, Rathkopf DE; COU-AA-302 Investigators. Abiraterone in metastatic prostate cancer without previous chemotherapy. N Engl J Med. 2013 Jan 10;368(2):138-48. doi: 10.1056/NEJMoa1209096. Epub 2012 Dec 10. PMID 23228172
- [Background] Rathkopf DE, Morris MJ, Fox JJ, Danila DC, Slovin SF, Hager JH, Rix PJ, Chow Maneval E, Chen I, Gonen M, Fleisher M, Larson SM, Sawyers CL, Scher HI. Phase I study of ARN-509, a novel antiandrogen, in the treatment of castration-resistant prostate cancer. J Clin Oncol. 2013 Oct 1;31(28):3525-30. doi: 10.1200/JCO.2013.50.1684. Epub 2013 Sep 3. PMID 24002508
- [Background] Clegg NJ, Wongvipat J, Joseph JD, Tran C, Ouk S, Dilhas A, Chen Y, Grillot K, Bischoff ED, Cai L, Aparicio A, Dorow S, Arora V, Shao G, Qian J, Zhao H, Yang G, Cao C, Sensintaffar J, Wasielewska T, Herbert MR, Bonnefous C, Darimont B, Scher HI, Smith-Jones P, Klang M, Smith ND, De Stanchina E, Wu N, Ouerfelli O, Rix PJ, Heyman RA, Jung ME, Sawyers CL, Hager JH. ARN-509: a novel antiandrogen for prostate cancer treatment. Cancer Res. 2012 Mar 15;72(6):1494-503. doi: 10.1158/0008-5472.CAN-11-3948. Epub 2012 Jan 20. PMID 22266222
- [Background] Rathkopf DE, Antonarakis ES, Shore ND, et al: ARN-509 in men with metastatic castration-resistant prostate cancer (mCRPC). J Clin Oncol 31:abstr 48, 2013
- [Background] Efstathiou E, Titus M, Wen S, Troncoso P, Hoang A, Corn P, Prokhorova I, Araujo J, Dmuchowski C, Melhem-Bertrandt A, Patil S, Logothetis CJ. Enzalutamide in Combination with Abiraterone Acetate in Bone Metastatic Castration-resistant Prostate Cancer Patients. Eur Urol Oncol. 2020 Feb;3(1):119-127. doi: 10.1016/j.euo.2019.01.008. Epub 2019 Apr 20. PMID 31412017
- [Background] Tombal B, Borre M, Rathenborg P, Werbrouck P, Van Poppel H, Heidenreich A, Iversen P, Braeckman J, Heracek J, Baskin-Bey E, Ouatas T, Perabo F, Phung D, Hirmand M, Smith MR. Enzalutamide monotherapy in hormone-naive prostate cancer: primary analysis of an open-label, single-arm, phase 2 study. Lancet Oncol. 2014 May;15(6):592-600. doi: 10.1016/S1470-2045(14)70129-9. Epub 2014 Apr 14. PMID 24739897
- [Derived] Bastos DA, Soares A, Schutz FAB, Cronemberger E, de Almeida Luz M, Martins SPDS, Muniz DQB, Carcano FM, Smaletz O, Peixoto FA, Gomes AJ, Cruz FM, Franke FA, Herchenhorn D, Gidekel R, Werutsky G, Rebelatto TF, Gomes de Jesus R, Souza VC, Fay AP, Maluf FC. Androgen Receptor Pathway Inhibitor Therapy for Advanced Prostate Cancer: Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Jan 2;8(1):e2454253. doi: 10.1001/jamanetworkopen.2024.54253. PMID 39804646
- [Derived] Maluf FC, Schutz FA, Cronemberger EH, Luz MA, Martins SPS, Muniz DQB, Bastos DA, Carcano FM, Smaletz O, Soares A, Peixoto FA, Gomes AJ, Cruz FM, Franke FA, Herchenhorn D, Dos Santos TM, Fabricio VC, Gidekel R, Werutsky G, de Jesus RG, Souza VC, Fay AP. A phase 2 randomized clinical trial of abiraterone plus ADT, apalutamide, or abiraterone and apalutamide in patients with advanced prostate cancer with non-castrate testosterone levels (LACOG 0415). Eur J Cancer. 2021 Nov;158:63-71. doi: 10.1016/j.ejca.2021.08.032. Epub 2021 Oct 13. PMID 34655838
- [Derived] Werutsky G, Maluf FC, Cronemberger EH, Carrera Souza V, Dos Santos Martins SP, Peixoto F, Smaletz O, Schutz F, Herchenhorn D, Santos T, Mavignier Carcano F, Queiroz Muniz D, Nunes Filho PRS, Zaffaroni F, Barrios C, Fay A. The LACOG-0415 phase II trial: abiraterone acetate and ADT versus apalutamide versus abiraterone acetate and apalutamide in patients with advanced prostate cancer with non-castration testosterone levels. BMC Cancer. 2019 May 23;19(1):487. doi: 10.1186/s12885-019-5709-y. PMID 31122212